CLINICAL TRIAL: NCT03292003
Title: Safety and Performance of Journey II BCS Total Knee System. A Retrospective, Multicenter Study
Brief Title: Journey II Bi-Cruciate Stabilized (BCS) Total Knee System Retrospective Study
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-4049-08
Record Dates: First submitted 2017-05-20; First posted 2017-09-25 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Total Knee Arthroplasty
Keywords: rheumatoid arthritis; post-traumatic arthritis; osteoarthritis; degenerative arthritis; failed osteotomy
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Journey II BCS Total Knee System: Subjects having TKA with Journey II BCS Total Knee System
  Interventions: Device: Journey II BCS Total Knee System

INTERVENTIONS:
Device: Journey II BCS Total Knee System

SUMMARY:
The objective of this study is to estimate the safety and performance of Journey II BCS TKS.

DETAILED DESCRIPTION:
The objective of this study is to estimate the safety and performance of Journey II BCS TKS. Specifically, the study will establish revision rate, treatment- and device-related complications, and clinical outcomes in a large sample of subjects who received the study device. Subjects are screened consecutively, beginning at the earliest date of implantation at each investigative site. Further, reasons for revision will be collected and analyzed. An analysis will be performed to identify characteristics (patient, surgeon and surgical) associated with an increased risk for revision. Finally, clinical, functional and quality of life outcomes will be analyzed to the extent data is available, given the retrospective study design.

ELIGIBILITY:
Inclusion Criteria:

* Subject received primary uni- or bi-lateral total knee arthroplasty with the Journey II BCS Total Knee System for approved indication
* The TKA occurred at least 12 weeks prior to enrollment
* Subject records contain Patient Reported Outcome data obtained ≤3 months prior to as well as ≥6 months post-enrollment.

Exclusion Criteria:

* Subject received the JOURNEY II BCS Total Knee System on the affected knee as a revision for a previously failed total or unicondylar knee arthroplasty

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sites will identify potential subjects by retrospectively reviewing their source documents in order to identify all patients who received TKA with the Journey II BCS TKS.
Sampling Method: Non-Probability Sample
Enrollment: 1694 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Revision Rate of Total Knee System | implantation through study completion, approximately 3 years
  Number of revisions

SECONDARY OUTCOMES:
Adverse Events | implantation through study completion, approximately 3 years
  Number of adverse events reported per ISO 14155 guidelines
Health care utilization: Hospitalization | implantation through study completion, approximately 3 years
  Length of hospital stay for primary (index) surgery
Health care utilization: Hospitalization | implantation through study completion, approximately 3 years
  Hospitalizations (admission for inpatient care) occurring after the hospitalization for the index surgery (number and length of stay)
Health care utilization: Rehabilitation | implantation through study completion, approximately 3 years
  number of sessions and duration of rehabilitation in weeks
Health care utilization: Outpatient visits | implantation through study completion, approximately 3 years
  Number and type of outpatient visits
Health Care Utilization: Re-operations | implantation through study completion, approximately 3 years
  number of re-operations and revisions
Patient reported outcomes | implantation through study completion, approximately 3 years
  EQ-5D-3L
Clinical outcomes | implantation through study completion, approximately 3 years
  Knee Society Score
Return to Work | implantation through study completion, approximately 3 years
  Changes in employment status will be recorded with the date on which the change occurred and the change status.
Technical Difficulties Encountered During Device Implantation | implantation through study completion, approximately 3 years
  Number of technical difficulties encountered with the device

CONTACTS AND LOCATIONS:
Overall Officials: Beate Hanson, MD, PhD, Study Chair — Vice President, Global Clinical Strategy
Locations (12):
- United States (9):
  - University of Colorado Orthopaedics, Aurora, Colorado
  - Andrews Research and Education Foundation, Gulf Breeze, Florida
  - Methodist Sports Medicine, Indianapolis, Indiana
  - Hospital for Special Surgery, New York, New York
  - University Orthopaedics Center, State College, Pennsylvania
  - TN Orthopaedic Foundation for Education and Research, Knoxville, Tennessee
  - San Antonio Orthopaedic Specialists, San Antonio, Texas
  - Providence Regional Medical Center, Everett, Washington
  - Marra Knee and Shoulder Center, Wheeling, West Virginia
- Belgium (2):
  - Jesse Ziekenhuis, Hasselt
  - UZ Leuven Campus, Pellenberg
- Christen Ortho AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No